CLINICAL TRIAL: NCT05310760
Title: Effectiveness of Vitamin C Supplementation in Infants and Children Suffering of Nutritional Rickets
Brief Title: Effectiveness of Vitamin C Supplementation in Treatment of Rickets
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Abdel Maksoud, Lecturer of Clinical and Chemical Pathology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-23-2021
Record Dates: First submitted 2022-01-31; First posted 2022-04-05 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Nutritional Rickets; Bone Turnover Rate Disorder
Keywords: Nutritional Rickets; Vitamin C; Rickets; Bone Turnover; Osteocalcin
MeSH Terms: conditions — Vitamin D Deficiency; Rickets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C receiving (Active Comparator): Therapeutic doses of Vitamin C are added to rachitic children treatment
  Interventions: Drug: Vit C
- Non Vitamin C receiving (No Intervention): The traditional treatment of nutritional rickets

INTERVENTIONS:
Drug: Vit C — Oral vitamin C (100 mg three times daily for one week then 100 mg once daily for 1-3 months)
  Arms: Vitamin C receiving

SUMMARY:
Effectiveness of therapeutic dose of vitamin C in infants and children with nutritional rickets as an adjuvant therapy with vitamin D and calcium The study is two armed Randomized Control Trial, to validate the role of Vit C supplementation on bone turnover infants and children with nutritional rickets.

DETAILED DESCRIPTION:
* Population of study & disease condition The study will include 88 infants and children with nutritional rickets
* Study setting:

The patients will be recruited from out-patient clinic of Cairo University Children's Hospital.

- Inclusion criteria: Any infant or child between 6 months and 3 years with nutritional rickets

* Exclusion criteria:

  1. Unwilling to participate in the study.
  2. Non nutritional causes of rickets as hypoparathyroidism, renal causes, chronic liver disease, and malabsorption.
  3. Children on vitamin C supplements above Recommended Daily allowance
* Methodology in details:
* History including age, sex, onset of manifestations, nutritional history, family history of similar condition, history of tetany or convulsion, motor development, drug intake, fractures, history of dentition, and manifestations of vitamin C deficiency (musculoskeletal pain, irritability, loss of appetite, petechiae, ecchymosis, gingival bleeding, alopecia, and poor wound healing) will be taken.
* Examination including anthropometric measurements, limb deformities, anterior fontanelle, cranial sutures, teeth, and gingival mucosa.
* Serum measurements of calcium, phosphorous, alkaline phosphate, Parathyroid hormone, and 25 hydroxy-vitamin D will be done at first visit then follow up of serum calcium, phosphorous and alkaline phosphatase after 4 and 12 weeks after starting the treatment.
* Radiological investigation in the form of anterior view X-ray of the knee that reveals the metaphysis end and epiphysis of the femur and tibia will be done at first visit and follow up after 4 weeks.
* Serum level of post treatment N-MID-osteocalcin detection (marker of bone turnover) [6] by ELIZA , Catalogue number E1499Hu Bioassay technology la laboratory England/China

The patient will be randomized 1:1 by computer randomization sequence into two groups (A, B). All patients will receive therapeutic dose of vitamin D (either single-day dose of 600,000 U or daily doses of 5000 U for 2-3 months) and oral elemental calcium according to Recommended Daily allowance . However, group A will receive oral vitamin C (100 mg three times daily for one week then 100 mg once daily for 1-3 months) in addition to the above-mentioned treatment.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis:

* Nutritional rickets in infants or children between 6 months and 3 years.
* Normal liver and kidney functions.
* The parents must be compliant to the clinic visits and the treatment doses.

Exclusion Criteria:

* Unwilling to participate in the study.
* Non nutritional causes of rickets as hypoparathyroidism, renal causes, chronic liver disease, and malabsorption.
* Children on vitamin C supplements above RDA.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of therapeutic doses of vitamin C in clinical finding of rickets | After 1 month stating the trial
  Measuring the clinical finding of rickets by history taking from parents (abnormal gait , delayed dentition, delayed milestones)
Effectiveness of therapeutic doses of vitamin C on anthropometric measures clinical finding of rickets | After 1 month stating the trial
  Measuring the anthropometric measures with correlation to the baseline ,these measures includes : Body mass index
Effectiveness of therapeutic doses of vitamin C in clinical signs of rickets | After 1 month stating the trial
  Examination to monitor the other symptoms of rickets including bone tenderness , bone deformities , hypotonia.
Laboratory follow up of rachitic children and infants | after 1 month from stating the trial
  Follow up calcium , phosphorus , parathyroid hormone, vitamin D and bone mineralization (serum MID-Osteocalcin by ELIZA
Radiological assessment after treatment for bone healing | after 1 month from stating the trial
  X-Ray of both knees , in A-P view to show metaphysis and epiphysis of both femur and tibia to assess the osteopenia, bone frying and bone cupping

SECONDARY OUTCOMES:
Effectiveness of therapeutic doses of vitamin C in clinical finding of rickets | after 3 month from stating the trial
  Measuring the clinical finding of rickets by history taking from parents (abnormal gait , delayed dentition, delayed milestones)
Effectiveness of therapeutic doses of vitamin C on anthropometric measures clinical finding of rickets | after 3 month from stating the trial
  Measuring the clinical finding of rickets by anthropometric measures with correlation to the baseline ,these measures includes : Body mass index
Effectiveness of therapeutic doses of vitamin C in clinical signs of rickets | after 3 month from stating the trial
  Examination to monitor the other symptoms of rickets including bone tenderness , bone deformities , hypotonia.
Laboratory follow up of rachitic children and infants | after 3 month from stating the trial
  Follow up calcium , phosphorus , parathyroid hormone, vitamin D and bone mineralization (serum MID-Osteocalcin by ELIZA.
Radiological assessment after treatment for bone healing | After 3 month from stating the trial
  X-Ray of both knees , in A-P view to show metaphysis and epiphysis of both femur and tibia to assess the osteopenia, bone frying and bone cupping

CONTACTS AND LOCATIONS:
Overall Officials: Fatina Fadel, Prof, Principal Investigator — Professor of Pediatrics Faculty of Medicine Cairo University
Locations (1):
- Cairo University Faculty of Medicine ,Abo elrish Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publishing